CLINICAL TRIAL: NCT02843334
Title: Study of the Prevalence of Fabry Disease in French Dialysis Patients
Acronym: FABRYDIAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0271
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Fabry Disease; End Stage Renal Disease; Renal Dialysis
Keywords: Fabry disease; End Stage Renal Disease; chronic dialysis; alpha galactosidase A; Lyso-GB3; GLA mutation; Prevalence
MeSH Terms: conditions — Fabry Disease; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood drops will be collected during a hemodialysis session and deposited on an anonymized blotting paper. Mutational analysis with sequencing of the whole GLA gene will be done to confirm the diagnosis of Fabry disease
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Population of adult patients undergoing chronic renal dialysis: Population of adult patients undergoing chronic renal dialysis for end stage kidney disease in 5 French areas (Rhône-Alpes-Auvergne, Ile de France, Aquitaine, Picardie and department of Gard)
  Interventions: Biological: Dried blood spot (DBS) sampling

INTERVENTIONS:
Biological: Dried blood spot (DBS) sampling — DBS be collected during a hemodialysis session and deposited on an anonymized blotting paper. Laboratory ARCHIMED Life Science GmbH, based in Austria will perform all the biological analysis. For the diagnosis, men will have a measure of the alpha-galactosidase activity level, whereas screening in women will be established on the association of alpha-galactosidase activity and lyso-GB3 analyses. If results are compatible, genetic mutation will be searches in order to confirm the diagnosis for women.

SUMMARY:
Fabry Disease (FD) is a rare genetic lysosomal storage disease including an X-linked mutation and characterized by an alpha-galactosidase A (GLA) deficiency. It causes globotriaosylceramide (GB3) accumulation within blood vessels, tissues and organs. This accumulation leads to multisystemic deficiency, such as progressive kidney insufficiency. Due to its low prevalence and non-specific symptoms, FD is under-diagnosed. Its estimated incidence is ranged from 1/40,000 to 1/120,000 live births. A review of the international literature suggests a higher prevalence among dialysis patients. Its diagnosis could lead to an enzyme replacement therapy, in order to avoid the occurrence or aggravation of other organs irreversible lesions, and to enhance the familial screening.

We aim to conduct a multicentric cross-sectional prevalence study in 5 areas (Rhône-Alpes-Auvergne, Ile de France, Aquitaine, Picardie and department of Gard), involving biologic collection and genetic diagnosis test. Our objective is to measure the prevalence of FD among dialysis patients. Eligible patients will be included after signing the informed consent.

In the five participating areas, all of the dialysis centers will be asked for involvement. Nominative data of the French renal epidemiology and information network (REIN) registry will enable first patients screening for eligibility among prevalent dialysis patients. If needed (insufficient or absent data in the REIN registry), data will be completed with medical files.

A blood drop will be collected during a hemodialysis session (or the monthly test for peritoneal dialysis treated patients) and deposited on an anonymized blotting paper. For the diagnosis of FD, men will have a measure of the alpha-galactosidase activity, whereas screening in women will be established on the association of alpha-galactosidase activity and lyso-GB3 analysis. If results are compatible with FD, genetic mutation will be search in order to confirm the diagnosis for women, and, for all, to offer familial testing. Results will be transmitted to the nephrologist within the next 2 to 9 weeks. Patients diagnosed with FD will be managed in accordance with the guidelines of the French National Authority for Health (F.N.A.H.).

ELIGIBILITY:
Inclusion Criteria:

* Woman or men
* Age between 18 to 70 years
* Patient undergoing chronic renal dialysis with a confirmed diagnosis of FD or a diagnosis of nephropathy according to the French renal epidemiology and information network (REIN) registry classification :
* Primitive glomerulonephritis
* Hypertension
* Diabetic nephropathy with non type 1 diabetes
* Vascular nephropathy
* Pyelonephritis
* Unknown or other
* Informed consent signed

Exclusion Criteria:

* IgA nephropathy confirmed by renal biopsy
* Diabetic nephropathy with type 1 diabetes
* Autosomal dominant polycystic kidney disease
* Law-protected patient
* Patient who doesn't belong to the national social security system, or similar system
* Pregnant or lactating woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of adult patients undergoing chronic renal dialysis for end stage kidney disease in 5 French areas (Rhône-Alpes-Auvergne, Ile de France, Aquitaine, Picardie and department of Gard)
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Fabry disease | during a hemodialysis session (Day 1)
  Analysis for the diagnostic of FD will be performed on blood drops:
  * For men : alpha galactosidase A enzyme activity (positive test if < 1,2µmol/L/h)
  * For women : alpha galactosidase A enzyme activity (positive test if < 1,2µmol/L/h) and lyso-GB3 (positive test if > 6 ng/mL) analysis. If results are compatible, GLA mutation will be confirmed by genotyping.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent JUILLARD, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (5):
- France (5):
  - Hôpital Pellegrin Tripode, Service de néphrologie-Dialyse, place Amélie Rabat Léon, Bordeaux, Aquitaine
  - Hôpital Universitaire Carémeau, Service de Néphrologie, Place du Pr R. Debré, Nîmes, Gard
  - CHU d'Amiens, Site Sud, Service de néphrologie, D408, Amiens, Nord Picardie
  - Hospices Civils de Lyon, Hôpital E Herriot, Service de néphrologie, 5 place d'Arsonval, Lyon, Rhones Alpes
  - Hôpital Necker, APHP Paris, Service de néphrologie-dialyse, 149 rue de Sèvres, Paris, Île-de-France Region